CLINICAL TRIAL: NCT04339426
Title: Open-Label, Non-Randomized Study to Evaluate Anti-Malarial/Anti-Infective Combination Therapies in Patients With Confirmed COVID-19 Infection
Brief Title: Atovaquone and Azithromycin Combination for Confirmed COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor enrollment
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRI-COVID-19-Anti-Malarial-001
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Atovaquone; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atovaquone/Azithromycin (Experimental): Atovaquone 750 mg PO Q12H for up to 10 days Azithromycin 500 mg PO Day 1 followed by 250 mg PO daily for up to 10 days (Days 2-10)
  Interventions: Drug: Atovaquone/Azithromycin

INTERVENTIONS:
Drug: Atovaquone/Azithromycin — Atovaquone 750 mg PO Q12H for up to 10 Days Azithromycin 500 mg PO Daily 1 followed by 250 mg PO Daily for up to 10 days (days 2-10)
  Other Names: Mepron/Zithromax

SUMMARY:
This study will evaluate anti-malarial/anti-infective single-agent and in combination for patients with confirmed COVID-19 infection. The first combination to be evaluated is atovaquone and azithromycin.

DETAILED DESCRIPTION:
This is an open-label, non-randomized study to evaluate anti-malarial/anti-infective single-agents and combination therapies for patients with confirmed COVID-19 infection requiring therapy as determined by risk factors for complication (age, comorbid illness) or the presence of respiratory compromise. The first combination to be evaluated is atovaquone/azithromycin. Other combinations may be added to the study at future amendments as information of potential benefit arises. The first part of the study will enroll 25 evaluable male and female patients 18 years of age or older with confirmed COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients age 18 years or older
* COVID-19 confirmed positive test results
* High risk for complications including with Medium (5-6) or High (More than or equal to 7) NEWS score
* Hematology criteria: ANC >500 cells/mcl, HGB >9 g/dl, Platelet count >75,000/mcl
* Metabolic criteria: Serum creatinine <2.0 mg/dl or calculated creatinine clearance (using Cockcroft-Gault) >30 ml/min, AST/ALT <5x ULN AND Total Bilirubin WNL (for patients with Gilbert's disease, direct bilirubin <ULN)

Exclusion Criteria:

* COVID-19 negative test result
* Inability to adhere to study protocol requirements
* Inability to provide informed consent
* Other acute or chronic medical or psychiatric condition that in the judgment of the investigator would make the participant inappropriate to take part in the study
* Pregnant and breastfeeding individuals
* QTc interval greater than 470 msecs at baseline
* History of hypersensitivity to atovaquone and/or azithromycin.
* History of known intolerance to atovaquone and/or azithromycin

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Virology Cure Rate | 10 days
  COVID-19 serology testing

SECONDARY OUTCOMES:
Incidence of GI adverse events | 47 days
  Measure incidence of diarrhea, vomiting, nausea and constipation
Cardiac Toxicity | 10 days
  12-Lead ECG daily if QTc >500 msec

OTHER OUTCOMES:
Changes in WBC w Diff, B cells, T cells, NK cells | 10 days
  Measure blood counts
Changes in cytokine levels, IL-1, IL-6, IL-12, IL-18, TNF-a | 10 days
  Measure changes in plasma cytokines throughout course of infection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gordon, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No